CLINICAL TRIAL: NCT00830310
Title: Customized Adherence Enhancement (CAE) Among Individuals With Bipolar Disorder
Brief Title: Customized Medication Adherence Enhancement for Adults With Bipolar Disorder
Acronym: UH CAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Martha Sajatovic, Professor of Psychiatry, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ-IRUSQUET0455; L1195
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Bipolar Disorder
Keywords: Patient Non-Adherence; Patient Non-Compliance; Patient Nonadherence; Patient Noncompliance; Patient Refusal of Treatment; Refusal of Treatment; Treatment Refusal
MeSH Terms: conditions — Bipolar Disorder; Patient Compliance; Treatment Refusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Customized Adherence Enhancement (CAE) (Experimental): Participants will be assigned to receive one or more of the study interventions based upon the participant's responses on the Attitudes toward Mood Stabilizers Questionnaire (AMSQ) and reasons for non-adherence on the Rating of Medication Influences (ROMI).
  Individuals will participate in a series of 4 60-minute sessions over a 4-week period, with the study therapist who will implement the module-based intervention. The number of modules may differ depending on the baseline adherence profile of the participant.
  An intervention manual developed by the investigators will provide explicit guidelines regarding how modules may be co-administered in single or multiple sessions to minimize redundancy as well as time and effort burden on study participants. The manual for each module will specifically address how any module could be combined with the other modules.
  Interventions: Behavioral: Psychoeducation module; Behavioral: Substance use module; Behavioral: Improved communication/rapport with provider module; Behavioral: Medication routines management module

INTERVENTIONS:
Behavioral: Psychoeducation module — Individuals will be assigned the psychoeducation module if they are identified as having opposition to prophylaxis, denial of illness severity or therapeutic effectiveness, negative attitudes towards drugs in general, or lack of information about mood stabilizers operationalized as a score of "1" or higher on any of these AMSQ subscales. Additionally, those individuals who are non-adherent/sub-optimally adherent because of stigma or embarrassment over medications or in relation to the use of complementary or alternative treatments will be assigned to participate in the psychoeducation module (ROMI stigma item or complementary/alternative treatment supplemental item).
Behavioral: Substance use module — Individuals will be assigned the substance use module if they endorse the ROMI substance use item or if substance use is identified as problematic on the clinician assessment.
Behavioral: Improved communication/rapport with provider module — Individuals will be assigned the provider communication/rapport module if they are identified as having fear of side effects operationalized as a score of "1" or higher on these AMSQ items. Additionally, those individuals who are non-adherent/suboptimally adherent because of concern regarding change in appearance "appearing medicated" or who experience side-effect-related distress as identified by the ROMI will be assigned the provider communication module.
Behavioral: Medication routines management module — Individuals will be assigned the medication routines management module if they are identified as having difficulties with medication routines operationalized as a score of "1" or higher on this AMSQ sub-scale, or if they are identified as experiencing outside opposition to medications by the ROMI.

SUMMARY:
This study is a modular intervention that is intended to improve treatment adherence among individuals with bipolar disorder on atypical antipsychotic therapy who have been identified as having treatment adherence problems.

DETAILED DESCRIPTION:
This study is a pilot, prospective project of the effects of customized adherence enhancement (CAE) when added to the medical management (usual care) of outpatients with bipolar disorder (BPD) who are patients at University Hospitals of Cleveland Case Medical Center, and who are known to be at risk for treatment non-adherence. In the proposed trial, CAE is supported by manuals delivered as a series of four modules whose use will be determined based upon an individual's identified treatment adherence vulnerabilities. The modules are components of a single, customized intervention. Although some participants may receive a different combination or number of modules, the participants are neither analyzed separately as a subpopulation nor compared as subpopulations. Therefore participants are all part of a solitary study arm. The effectiveness of the entire customized intervention system is of interest.

All individuals will continue to receive treatment as usual with their regular provider. Those who are enrolled in the study intervention will participate in a series of 4 in-person meetings with the study interventionist over a 4-week time period and 1-2 telephone follow-ups. These meetings with the interventionist will consist of whatever modules were assigned at baseline that are customized to that particular participant's treatment adherence vulnerabilities. A total of 3 to 4 assessment meetings with the research assistant will occur over a three-month time period.

Primary objective The aim of this project is to test the use of a modular-based intervention in a pilot feasibility, acceptability and preliminary efficacy study of customized adherence enhancement (CAE) in a vulnerable population with BPD. We hypothesize that CAE will be: 1) feasible to administer within a academic medical center; 2) acceptable to participants with BPD; and 3) associated with improvements in treatment adherence.

Secondary objectives Individuals who receive CAE will have improvements in BPD symptoms, global psychopathology, overall treatment attitudes and in functional status.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Bipolar Disorder (BPD) Type I or Type II determined by a standardized diagnostic interview, the Mini-International Neuropsychiatric Interview (MINI) (Sheehan 1998);
* Demonstrated history of poor adherence as per either self-report or clinician report. In this study, self-reported treatment non-adherence will be identified with Tablet Routines Questionnaire (TRQ). Poorly adherent individuals will be defined as those who miss 20% or more of medication within either the past week or past month (those missing 20% or more within past week will be considered to be non-adherent over the past month).
* BPD for at least two years duration;
* Treatment with atypical antipsychotic medication to stabilize mood for at least six months;
* The ability to participate in psychiatric interviews and to give written, informed consent for study participation; and
* Age 18 or older.

Exclusion Criteria:

* Unable/unwilling to participate in psychiatric interviews based on the clinical opinion of the investigator or the treating clinician. Individuals who are grossly psychotic may be excluded at this point if the treating clinician feels that the prospective participant is unable to participate in the interviews or study procedures;
* Unable/unwilling to give written, informed consent to study participation;
* High risk for suicide (e.g., active suicidal ideation and recent suicide attempt; active suicidal ideation and current intent or plan). In the interest of patient safety, individuals who are acutely suicidal will be excluded from study participation; or
* Individuals who are non-English speaking will be excluded as study assessment tools are not available in other languages and would be impractical to develop in this small, exploratory study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University and University Hospitals Case Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in January of 2009 and the last participant was enrolled in June of 2010.
Groups:
- Customized Adherence Enhancement (CAE): Participants will be assigned to receive one or more of the study interventions based upon the participant's responses on the AMSQ and reasons for non-adherence on the ROMI.
  Individuals will participate in a series of 4 60-minute sessions over a 4-week period, with the study therapist who will implement the module-based intervention. The number of modules may differ depending on the baseline adherence profile of the participant.
  An intervention manual developed by the investigators will provide explicit guidelines regarding how modules may be co-administered in single or multiple sessions to minimize redundancy as well as time and effort burden on study participants. The manual for each module will specifically address how any module could be combined with the other modules.
Period: Overall Study
Arm/Group | Customized Adherence Enhancement (CAE)
Started | 43
Completed | 30
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Change in Treatment Non-adherence as Measured by the Tablets Routine Questionnaire (TRQ) (Past Month)
Description: Treatment non-adherence is measured as a percentage of medications not taken within the past month at time of assessment.
  The minimum score is 0 and the maximum score is 100. A higher score implies poorer treatment adherence.
Time Frame: From Baseline to 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: percentage of medication not taken
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
percentage of medication not taken | -23.6 (4.5)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 3 months and baseline equals zero; Test type: Superiority or Other; p < 0.001, Sign test

2. Secondary Outcome: Change in Symptoms of Bipolar Disorder as Measured by the Young Mania Rating Scale (YMRS)
Description: The minimum possible score is 0 and the maximum score is 60. A higher score implies a worse condition.
Time Frame: From Baseline to 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 29
units on a scale | -3.7 (1.1)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = 0.002, Sign test

3. Secondary Outcome: Change in Global Psychopathology as Measured by the Clinical Global Impression Scale (CGI)
Description: The minimum possible score is 1 and the maximum score is 7. A higher score implies a worse condition.
Time Frame: From Baseline to 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
units on a scale | -0.67 (0.18)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

4. Secondary Outcome: Change in Overall Treatment Attitudes as Measured by the Drug Attitude Inventory (DAI)
Description: The minimum score is 0 and the maximum score is 10. A higher score implies a better attitude.
Time Frame: From Baseline to 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
units on a scale | 1.7 (0.46)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

5. Secondary Outcome: Change in Functional Status as Measure by the Global Assessment of Functioning Scale (GAF)
Description: The minimum score is 1 and the maximum score is 100. A higher score implies higher functioning.
Time Frame: From Baseline to 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 29
units on a scale | 8.2 (2.2)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = 0.001, Sign test

6. Secondary Outcome: Change in Symptoms of Bipolar Disorder as Measured by the Hamilton Depression Rating Scale (HAM-D)
Description: The minimum score is 0 and the maximum score is 52. A higher score implies a worse condition.
Time Frame: From Baseline to 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 29
units on a scale | -2.4 (0.88)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = 0.011, t-test, 2 sided

7. Secondary Outcome: Change in Symptoms of Bipolar Disorder as Measured by the Brief Psychiatric Rating Scale (BPRS)
Description: The minimum score is 18 and the maximum score is 126. A higher score implies a worse condition.
Time Frame: From Baseline to 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 29
units on a scale | -3.4 (1.5)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = 0.038, t-test, 2 sided

8. Primary Outcome: Change in Treatment Non-adherence as Measured by the Tablets Routine Questionnaire (TRQ) (Past Week)
Description: Treatment nonadherence is measured as a percentage of medications not taken within the past week at time of assessment.
  The minimum score is 0 and the maximum score is 100. A higher score implies poorer treatment adherence.
Time Frame: From Baseline to 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: percentage of medications not taken
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
percentage of medications not taken | -17.8 (5.7)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the median difference between 3 months and baseline equals zero; Test type: Superiority or Other; p = 0.002, Sign test

9. Primary Outcome: Change in Treatment Adherence as Measured by the Morisky Scale
Description: The minimum score is 0 and the maximum score is 4. A higher score implies poorer treatment adherence.
Time Frame: From Baseline to 3 months
Population: Number of participants for analysis was based on all available data at the three month time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Customized Adherence Enhancement (CAE)
Number analyzed (Participants) | 30
units on a scale | -1.4 (0.32)
Statistical Analysis 1: Comparison: Customized Adherence Enhancement (CAE); The null hypothesis is that the mean difference between 3 months and baseline equals zero; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Customized Adherence Enhancement (CAE)
Serious Adverse Events (participants affected / at risk) | 4/43
Other Adverse Events (participants affected / at risk) | 1/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Customized Adherence Enhancement (CAE) (N=43)
broken vertebrae (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant was in a car accident and received a broken vertebrae
worsening depression (Psychiatric disorders) | 1 (1) — Participant hospitalized for worsening depression
congestive heart failure (Cardiac disorders) | 1 (1) — Participant was hospitalized and diagnosed with congestive heart failure
worsening mania (Psychiatric disorders) | 1 (2) — Participant took more medication than prescribed hoping to treat their mania and was hospitalized
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Customized Adherence Enhancement (CAE) (N=43)
substance abuse (Psychiatric disorders) | 1 (1) — Subject caused a car accident while drunk driving

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days